CLINICAL TRIAL: NCT02536495
Title: An Investigator-Sponsored Phase 1/2 Study of Selinexor (KPT-330) and Docetaxel as Second Line Therapy in Patients With Relapsed Squamous Cell Lung Cancer
Brief Title: Selinexor and Docetaxel in Treating Patients With Recurrent or Metastatic Squamous Cell Lung Cancer
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: PI decision due to funding support
Sponsor: Erin Bertino (Other)
Collaborators: Karyopharm Therapeutics Inc (Industry)
Responsible Party: Sponsor-Investigator, Erin Bertino, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-14152; NCI-2015-01165 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2015-08-27; First posted 2015-09-01 (Estimated); Last update posted 2015-10-30 (Estimated); Status verified 2015-10

CONDITIONS: Recurrent Squamous Cell Lung Carcinoma; Stage IV Squamous Cell Lung Carcinoma
MeSH Terms: interventions — Docetaxel; selinexor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (docetaxel, selinexor) (Experimental): Patients receive docetaxel IV on day 1 and selinexor PO BID on days 1, 3, 7, 9, 13, and 15. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Docetaxel; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Selinexor

INTERVENTIONS:
Drug: Docetaxel — Given IV
  Other Names: RP56976; Taxotere; Taxotere Injection Concentrate
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Drug: Selinexor — Given PO
  Other Names: CRM1 Nuclear Export Inhibitor KPT-330; KPT-330; Selective Inhibitor of Nuclear Export KPT-330; SINE KPT-330

SUMMARY:
This phase I/II trial studies the side effects and best dose of selinexor and docetaxel and to see how well they work when given together in treating patients with squamous cell lung cancer that has come back or spread to other places in the body. Selinexor may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving selinexor together with docetaxel may work better in treating squamous cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the toxicity and determine recommended phase II dose of the combination of docetaxel and selinexor. (Phase I) II. To evaluate the efficacy as measured by progression free survival (PFS) of docetaxel and selinexor in patients with recurrent/metastatic squamous cell lung cancer. (Phase I/II)

SECONDARY OBJECTIVES:

I. To evaluate the objective tumor response rate as determined by radiographic response.

II. To evaluated the disease control rate (complete response, partial responses, and stable disease).

III. To evaluate the overall survival (OS). IV. To evaluate the safety and tolerability of single agent selinexor.

TERTIARY OBJECTIVES:

I. Lung cancer genomics sequencing panel. II. Tumor biopsy (baseline and cycle 2). III. Plasma cytokine analysis, peripheral blood ribonucleic acid (RNA) analysis.

OUTLINE: This is a phase I, dose-escalation study followed by a phase II study.

Patients receive docetaxel intravenously (IV) on day 1 and selinexor orally (PO) twice daily (BID) on days 1, 3, 7, 9, 13, and 15. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up monthly for 3 months, every 3 months for 9 months, and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent in accordance with federal, local, and institutional guidelines
* Patients with recurrent or metastatic squamous cell carcinoma of the lung - diagnosis must be histologically confirmed
* Measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST 1.1) at the time of study entry
* Objective evidence of disease progression on study entry
* Prior systemic anticancer therapy: Patients will have received at least 1 platinum-based chemotherapy regimen, but no more than 2 cytotoxic chemotherapy regimens in the setting of recurrent or metastatic disease; the regimen(s) may have included biological, molecularly targeted or immune therapies; adjuvant chemotherapy is considered 1 cytotoxic chemotherapy regimen if the last administration occurred < 1 year prior to entry
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Absolute neutrophil count (ANC) > 1500/mm^3
* Platelets count > 100,000 mm^3 and less than 1,000,000 mm^3
* Total bilirubin < 2 times the upper limit of normal (ULN) (except patients with Gilbert's syndrome who must have a total bilirubin of < 3 times ULN)
* Alanine aminotransferase (ALT) < 2.5 times ULN; in the case of known (radiological and/or biopsy documented) liver metastasis, ALT < 5.0 times ULN is acceptable; patients with > 3 liver metastases at enrollment will be excluded
* Estimated creatinine clearance of >= 30 mL/min, calculated using the formula of Cockcroft and Gault
* Amylase =< 1.5 x ULN
* Lipase =< 1.5 x ULN
* Alkaline phosphatase limit =< 2.5 x ULN
* Female patients of child-bearing potential must agree to use dual methods of contraception and have a negative serum pregnancy test at screening; male patients must use an effective barrier method of contraception if sexually active with a female of child-bearing potential throughout the study and for three months following the last dose of selinexor
* Resolution to grade =< 1 by National Cancer Institute Common Terminology Criteria for Adverse Events version 4.03 (CTCAE v4.03) of all clinically significant toxic effects of prior anti-cancer therapy (with the exception neuropathy, which may be =< grade 2 within 14 days prior to cycle 1 day 1)

Exclusion Criteria:

* Patients who are pregnant or lactating
* Radiation, chemotherapy, or immunotherapy or any other anticancer therapy =< 2 weeks prior to cycle 1 day 1
* Prior treatment with selective inhibitor of nuclear export (SINE) inhibitor
* Major surgery within four weeks before cycle 1, day 1
* Unstable cardiovascular function:

  * Electrocardiography (ECG) abnormalities requiring treatment, or
  * Congestive heart failure (CHF) of New York Heart Association (NYHA) class >= 3
  * Myocardial infarction (MI) within 3 months
* Uncontrolled infection requiring parenteral antibiotics, antivirals, or antifungals within one week prior to first dose; patients with controlled infection or on prophylactic antibiotics are permitted in the study
* Known to be human immunodeficiency virus (HIV) seropositive
* Known active hepatitis A, B, or C infection; or known to be positive for hepatitis C virus (HCV) RNA or hepatitis B surface antigen (HBsAg) (hepatitis B virus [HBV] surface antigen)
* Any underlying condition that would significantly interfere with the absorption of an oral medication
* Patients with markedly decreased visual acuity
* Serious psychiatric or medical conditions that could interfere with treatment
* Participation in an investigational anti-cancer study =< 3 weeks prior to cycle day 1
* Concurrent therapy with approved or investigational anticancer therapeutic other than steroids
* Patients with coagulation problems and active bleeding in the last month (peptic ulcer, epistaxis, spontaneous bleeding)
* Uncontrolled brain metastases; patients with brain metastases are permitted if they have received appropriate therapy and demonstrated control of the brain metastases following therapy; patients with known brain metastases will require magnetic resonance imaging (MRI) brain to demonstrate disease control prior to enrollment (lack of symptom progression for two weeks off therapeutic doses of steroids, excluding chronic steroids used for control of chronic obstructive pulmonary disease [COPD])
* Renal failure requiring hemodialysis or peritoneal dialysis
* Patients with significantly diseased or obstructed gastrointestinal tract, malabsorption, uncontrolled vomiting or diarrhea or inability to swallow oral medications
* Patients who are severely underweight in the opinion of the investigator
* Prior cancer diagnosis is allowed if patient is disease-free for >= 3 years, or disease free for < 3 years for treated basal cell/squamous cell skin cancer or in situ cervical cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-09; Primary Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | Time from the date of study registration to the date of disease progression or to the date of last observation when no event (disease progression) has occurred, assessed up to 3 years
  PFS will be estimated by the method of Kaplan and Meier (KM). Appropriate one-sided 90% confidence boundary will also be calculated for the final test KM test statistic at 12 weeks.

SECONDARY OUTCOMES:
Disease control rate (Complete Response + Partial Response + stable disease) | Up to 1 year
  An analysis of disease control rate will be performed. These estimates will be accompanied by exact binomial confidence intervals as well.
Incidence of adverse events, graded according to the National Cancer Institute CTCAE version 4.03 | Up to 1 year
  Frequency and severity of adverse events and tolerability of the regimen will be collected and summarized by descriptive statistics for each of the disease cohorts. The maximum grade for each type of toxicity will be recorded for each patient, and frequency tables will be reviewed to determine toxicity patterns.
Objective response rate (complete response [CR] or partial response [PR] by RECIST) | Up to 1 year
  Those who achieve PR or CR will be considered responses and the overall response rate will be calculated as the number of PRs and CRs divided by the total number of evaluable patients. These estimates will be accompanied by exact binomial confidence intervals as well.
Overall survival | Date of study registration to the date of event (i.e., death) or the date of last follow-up if no event has occurred at their last evaluation, assessed up to 3 years
  Kaplan-Meier curves will be used to estimate overall survival. Cox proportional hazards models will be further considered to explore a limited set of confounding factors.

OTHER OUTCOMES:
Changes in tumor suppressor protein expression levels | Baseline to up to course 2, day 1
  Tumor biopsies before and after therapy will be evaluated to assess baseline expression of tumor suppressor proteins and how change in these proteins may correspond with clinical outcomes of interest. Markers will be summarized by descriptive statistics overall and through stratified Kaplan Meier plots to explore differences in PFS. Generalized linear models will model changes in expression levels over time, with potential adjustment for confounding variables.

CONTACTS AND LOCATIONS:
Overall Officials: Erin Bertino, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu